CLINICAL TRIAL: NCT03415503
Title: Anthocyanin Supplementation Improves Blood Lipids in a Dose-response Manner in Subjects With Dyslipidemia
Brief Title: Dietary Anthocyanins Improve Lipid Metabolism in a Dose - Dependent Manner
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhanghy, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: lingwh87331597
Record Dates: First submitted 2017-12-12; First posted 2018-01-30 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Dyslipidemias
Keywords: anthocyanins; dyslipidemias; dose response
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- placebo (Placebo Comparator): The placebo capsules only contained pullulan and maltodextrin.During the trial period, the participants were instructed to consume 2 Medox® placebo capsules twice daily (30 min after breakfast or supper).
  Interventions: Drug: Medox® Anthocyanin capsules
- 40mg/d anthocyanins (Experimental): Medox® Anthocyanin capsules is consisted of 17 different natural purified anthocyanins.from bilberry (Vaccinium myrtillus) and black currant (Ribesnigrum). To achieve the double-blind,every group are instructed to consume the same amount of capsule. During the trial period, the participants will be instructed to consume one Medox® anthocyanin capsules and one Medox® placebo capsules 30 min after breakfast and consume two Medox® placebo capsules 30 min after supper.The anthocyanin capsules (40 mg anthocyanins per capsule) will provid a total daily intake of 40 mg anthocyanins.
  Interventions: Drug: Medox® Anthocyanin capsules
- 80mg/d anthocyanins (Experimental): Medox® Anthocyanin capsules is consisted of 17 different natural purified anthocyanins.from bilberry (Vaccinium myrtillus) and black currant (Ribesnigrum).To achieve the double-blind,every group are instructed to consume the same amount of capsule. During the trial period, the participants will be instructed to consume one Medox® anthocyanin capsules and one Medox® placebo capsules 30 min after breakfast and consume two Medox® placebo capsules 30 min after supper.The anthocyanin capsules (80 mg anthocyanins per capsule) will provid a total daily intake of 80 mg anthocyanins.
  Interventions: Drug: Medox® Anthocyanin capsules
- 320mg/d anthocyanins (Experimental): Medox® Anthocyanin capsules is consisted of 17 different natural purified anthocyanins.from bilberry (Vaccinium myrtillus) and black currant (Ribesnigrum).To achieve the double-blind,every group are instructed to consume the same amount of capsule. During the trial period, the participants will be instructed to consume two Medox® anthocyanin capsules 30 min after breakfast and after supper.The anthocyanin capsules (80 mg anthocyanins per capsule,4 per day) will provid a total daily intake of 320 mg anthocyanins.
  Interventions: Drug: Medox® Anthocyanin capsules

INTERVENTIONS:
Drug: Medox® Anthocyanin capsules — Subjects were orally administered Medox® capsules daily for 12 weeks.
  Other Names: Medox® Placebo capsules

SUMMARY:
In order to study the effect of anthocyanins on the improvement of glucose and lipid metabolism, randomized intervention trials were conducted to compare the effects of anthocyanins on the improvement of glucose and lipid metabolism in different dose groups.To explore the best dose of anthocyanins for the prevention and treatment of anthocyanin metabolic diseases provide an important scientific basis.

DETAILED DESCRIPTION:
In order to study the effect of anthocyanins on the improvement of glucose and lipid metabolism, randomized controlled trials were conducted to enrolled 300 patients with dyslipidemia. The subjects were divided into 0 mg / d, 40 mg / d, 80 mg / d, 320 mg/ d five dose groups, intervention for 12 weeks, comparing different doses of anthocyanins on glucose and lipid metabolism.To explore the best dose of anthocyanins for the prevention and treatment of anthocyanin metabolic diseases provide an important scientific basis.

ELIGIBILITY:
Inclusion Criteria:

* Dyslipidemia
* Subjects with dyslipidemia who also have prediabetes
* The age between 35 and 70 years old

Exclusion Criteria:

* intake of any medicine that affect lipid and glucose metabolism currently or in the preceding 6 months
* dietary supplementation with phytochemicals including anthocyanins in the preceding 2 months
* history of acute or chronic infectious disease, autoimmune disease, cancer, traumatic injury, or surgery in the preceding 1 month
* history of severe chronic disease including AS and CVD, liver or renal dysfunction, and lactation or pregnancy
* Pregnant woman and Breast Feeding Women

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Anthocyanins dose-dependently improved blood lipids in patients with dyslipidemia. | 12 weeks
  After 12 weeks intervention of anthocyanins, serum lipid profiles were measured at baseline, at 6 weeks, and at the end of 12 weeks.

SECONDARY OUTCOMES:
Anthocyanin supplementation improves cholesterol efflux capacity in a dose-response manner in subjects with dyslipidemia | 12 weeks
  After 12 weeks intervention of anthocyanins,cholesterol efflux capacity (CEC) were measured at baseline, at 6 weeks, and at the end of 12 weeks.
Anthocyanins supplementation improve anti-oxidative and anti-inflammation capacity in a dose-response manner in subjects with dyslipidemia. | 12 weeks
  After 12 weeks intervention of anthocyanins,Urine 8-iso-prostaglandinF2α (8-iso-PGF2α), 8-hydroxy-2'-deoxyguanosine (8-OHdG) and serum malondialdehyde (MDA), superoxide dismutase (SOD), UA (urine acid), interleukin-6 (IL-6), interleukin-10(IL-10), tumor necrosis factor-α (TNF-α) and C-reactive protein (CRP) were measured at baseline, at 6 weeks and at the end of 12 weeks.
Anthocyanins supplementation attenuate platelet hyperreactivity in a dose-response manner in subjects with dyslipidemia. | 12 weeks
  After 12 weeks intervention of anthocyanins, platelet aggregation, the expression of P-selectin (CD62p) activated GPⅡbⅢa (PAC-1), platelet reactive oxygen species (ROS) and platelet mitochondrial membrane potential (TMRM) were measured at baseline, at 6 weeks and at the end of 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ling W H, Pro, Study Chair — Department of Nutrition and Food Hygiene,School of Public Health, Sun Yat-sen University
Locations (1):
- Department of Nutrition and Food Hygiene,School of Public Health, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao Y, Xu H, Tian Z, Wang X, Xu L, Li K, Gao X, Fan D, Ma X, Ling W, Yang Y. Dose-dependent reductions in plasma ceramides after anthocyanin supplementation are associated with improvements in plasma lipids and cholesterol efflux capacity in dyslipidemia: A randomized controlled trial. Clin Nutr. 2021 Apr;40(4):1871-1878. doi: 10.1016/j.clnu.2020.10.014. Epub 2020 Oct 15. PMID 33131908